CLINICAL TRIAL: NCT01713829
Title: Cranberry Consumption Improves γδ T Cell Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: The Cranberry Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CB-472-2012
Record Dates: First submitted 2012-09-18; First posted 2012-10-25 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
Keywords: cranberry; gamma delta T cell; improvement in immune cell function in healthy humans; proliferation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cranberry Beverage (Experimental): Cranberry Beverage is provided in an 8 oz daily beverage consumed once daily for 12 weeks
  Interventions: Other: Cranberry Beverage
- Placebo Beverage (Placebo Comparator): The placebo beverage looks like the active arm and is given in the same way but contains no active ingredient.
  Interventions: Other: Placebo Beverage

INTERVENTIONS:
Other: Cranberry Beverage — 8 oz cranberry beverage consumed daily for 12 weeks
  Arms: Cranberry Beverage
Other: Placebo Beverage — 8 oz placebo beverage consumed daily for 12 weeks
  Arms: Placebo Beverage

SUMMARY:
The purpose of this study is to determine the extent to which consuming a cranberry beverage modifies immune function, specifically related to γδ T cells and other innate immune cells. It is hypothesized that cranberry components will interact with immune cells to activate signaling pathways that enhance cell function. Enhanced immune cell function should result in reduced number, duration, and severity of cold and flu symptoms.

ELIGIBILITY:
Inclusion Criteria:

* between 21 and 35 years of age and in good health
* have a BMI between 18.5 and 29.9
* willing to consume the study beverage for 12 weeks
* willing to have a small amount of blood drawn two times
* willing to stop consuming tea and immune-enhancing dietary supplements (e.g. antioxidant-, probiotic-, or flavonoid-containing supplements, fish oil, and Echinacea) before and during the 12 weeks of the study
* willing to consume no more than 7 servings of fruits and vegetables a day
* willing to limit your alcohol consumption to no more than 14 glasses a week
* willing to limit your yogurt consumption to no more than one 8oz. serving per day

Exclusion Criteria:

* have food allergies
* have hypertension
* taking non-steroidal anti-inflammatory drugs on a chronic basis, antibiotics, or immunosuppressive drugs
* sensitive to aspirin or prone to kidney stones
* current smoker
* pregnant, lactating, or on hormone therapy, except for birth control pills

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in Immune Cell Function | Measured at baseline and 6 weeks
  * Change in leukocyte phenotype
  * Change in the ability of the natural killer and/or γδ T cells to proliferate when cultured ex vivo
  * Change in peripheral blood mononuclear cell cytokine and chemokine production in response to mitogens

SECONDARY OUTCOMES:
Cold and Flu Symptoms | 12 weeks
  Incidence and severity of cold and flu symptoms, total and individual. Other signs of severity, for example, visits to doctor or health clinic, reduction in daily activities, prescribed or over-the-counter medications taken.

CONTACTS AND LOCATIONS:
Overall Officials: Susan S Percival, PhD, Principal Investigator — University of Florida
Locations (1):
- 449 Food Science and Human Nutrition Department, University of Florida, Gainesville, Florida, United States